CLINICAL TRIAL: NCT06718426
Title: Evaluation of Fertitonex Effects on Semen Parameters in Clinical Varicocele Patient, Placebo Controlled Study
Brief Title: Evaluation of Fertitonex Effects on Semen Parameters in Clinical Varicocele Patient.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fertitonex in varicocele
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Varicocele
Keywords: varicocele; Fertitonex; infertility; semen analysis
MeSH Terms: conditions — Varicocele; Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fertitonex group (Active Comparator): Patients in this group will receive Fertitonex which contains L- carnitine L-tartarate 300 mg, L-arginine 241mg, vitamin B6 1.1 mg, vitamin B12 1.7 mcg, vitamin D3 2 mcg, vitamin E 6.5 mg, vitamin C 60 mg, selenium 28 mcg, zinc 7.5 mg, folic acid 300 mcg and CoQ 10 enzyme 7.5 mg in each capsule. The dose will be one capsule twice daily for 3 months.
  Interventions: Drug: Fertitonex capsule
- Placebo group (Placebo Comparator): Patients in this group will receive placebo capsule twice daily for 3 months.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Fertitonex capsule — Fertitonex which contains L- carnitine L-tartarate 300 mg, L-arginine 241mg, vitamin B6 1.1 mg, vitamin B12 1.7 mcg, vitamin D3 2 mcg, vitamin E 6.5 mg, vitamin C 60 mg, selenium 28 mcg, zinc 7.5 mg, folic acid 300 mcg and CoQ 10 enzyme 7.5 mg in each capsule. The dose will be one capsule twice daily for 3 months.
  Arms: Fertitonex group
Drug: Placebo Oral Capsule — placebo oral capsule. the dose is twice daily for 3 months
  Arms: Placebo group

SUMMARY:
The aim of the study is to evaluate the Fertitonex effects on semen parameters in clinical varicocele patients.

DETAILED DESCRIPTION:
Infertility is defined as the inability of a couple to conceive after one year of unprotected, frequent and regular sexual intercourse. Almost 15% of all couples trying to conceive are affected by infertility, and in almost half of these cases male infertility is the sole or a contributing factor. The most common cause is idiopathic oligoasthenoteratozoospermia (OAT) that is defined as follows sperm concentration, the proportion of morphologically normal sperm and the proportion of motile sperm are all lower than the World Health Organization (WHO) reference values.

Despite extensive research, a successful treatment for OAT had not yet been developed. Small amounts of reactive oxygen species (ROS) are produced by spermatozoa in physiological conditions, and various scavengers act to reduce the concentration of these ROS in the seminal plasma. ROS are needed for capacitation, acrosome reaction and ultimately fertilization.

Antioxidants might help maintain the balance between ROS production and clearance and thus could improve sperm quality Additionally, observational studies had found a lower frequency of sperm aneuploidy in men with a higher dietary intake of antioxidants than in those with a lower intake. In semen, antioxidants decrease OS, potentially improving sperm motility and reducing DNA fragmentation.

We aim to evaluate the Fertitonex effects on semen parameters in clinical varicocele patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary infertility.
* Abnormal semen analysis parameters.
* Clinically evident varicocele confirmed by scrotal duplex.

Exclusion Criteria:

* 2ry infertility.
* Normal semen analysis parameters.
* Clinically non-evident varicocele.
* Past history of varicocelectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Total sperm count | 3 months
  Total sperm count will be assessed by Semen analysis done after 3 months of either fertitonex or placebo administration.
  Total sperm count will be measured by number of sperms present in the semen sample.
Sperm motility | 3 months
  Sperm motility will be assessed by semen analysis done after 3 months of either fertitonex or placebo administration.
  Both total motility will be measured by percentage of motile sperms and progressive motility will be measured by percentage of progressively motile sperms present in the semen sample.
Sperm Morphology | 3 months
  Sperm morphology will be assessed by semen analysis done after 3 months of either fertitonex or placebo administration.
  Sperm morphology will be measured by percentage of normally shaped sperms present in the semen sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt